CLINICAL TRIAL: NCT00698919
Title: Bacterial DNA Detection as a Diagnostic Tool of Infection in Critical Ill Patients With SIRS
Brief Title: Bacterial Infection Diagnosis Using Blood DNA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Delafontaine Hospital (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other); Jacques Cartier Institute (Unknown); Unity Health Toronto (Other); Institut Pasteur (Industry)
Responsible Party: Christophe Adrie, MD, PhD, RER Saint Denis
Other Study IDs: RCB : 2008-A00361-54; PF01743
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Infection; Sepsis
Keywords: Bacterial DNA; Systemic inflammatory response syndrome; Infection; Intensive Care Unit
MeSH Terms: conditions — Infections; Sepsis; Systemic Inflammatory Response Syndrome | interventions — Observation

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sample with bacterial DNA (and no human DNA will be studied)
  We will have also some blood and plasma for cytokines,peptidoglycan and endotoxin measurement.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Development cohort: A first group of one hundred patients with SIRS will be included to evaluate the accuracy of this new test.
  Interventions: Other: Observational study
- Validation Cohort: Depending on the result of the previous (development) cohort we will more accurately evaluate the need of number of patients with SIRS to include in the second cohort of patients.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is not an interventional studies. We will just compare two methods of bacterial diagnosis. Of note the physicians will care of their patients with the classic bacterial analysis tools; so there is no modification of the care.
  The new techniques used (DNA detection) will done later on and thus won't modify their decision.

SUMMARY:
Sepsis is a common cause of morbidity and death in intensive care units. Clinical and laboratory signs of systemic inflammation, including changes in body temperature, tachycardia, or leukocytosis, are neither sensitive nor specific enough for the diagnosis of sepsis. The diagnosis of sepsis is difficult, because clinical signs are unspecific. These signs include tachycardia, leucocytosis, tachypnoea, and pyrexia, which are collectively termed a systemic inflammatory response syndrome (SIRS). SIRS is very common in critically ill patients, being found in various conditions including trauma, surgery, burns, pancreatitis, post-cardiac arrest syndrome, cardiac surgery. Microbiological culture can be used to distinguish sepsis from non-infectious conditions. However, this method lacks sensitivity and specificity, and there is often a substantial time delay. So these signs can also be misleading because critically ill patients often present with the systemic inflammatory response syndrome without infection. This issue is of paramount importance, since therapy and outcome differ greatly between patients with and those without sepsis; clinicians are often prone to overuse antibiotic therapy being afraid of not treating a potential infection or superinfection. Moreover, the widespread use of antibiotics for all such patients is likely to increase antibiotic resistance, toxicity, and costs. On the opposite, any delay in administration of antibiotics can be extremely detrimental for the infected patient with an exponential increase of the odd ratio for death. Search for early biomarker tools for the diagnosis of infection, initially promising, are quite challenged and controversial nowadays because they can be more related to the inflammation response, irrespective to the insult. Furthermore up to 40% of the infections remain strongly suspected but not bacteriologically documented. Persisting researches are ongoing to find new markers to better discriminate SIRS related to infection process from to SIRS not related to infection. Cytokine profiles using multiplex analysis seems more related to the severity of the SIRS than the trigger of the SIRS (infectious or non infectious diseases). Thus, new tools have been developed to identify bacteria by detecting their DNA by various techniques. These techniques have many potential interests over conventional microbiologic tests by decreasing turnaround time (within a few hours 2-6 hours), reducing inhibitory effects of prior use of antibiotics, detection of slow or fastidious growing organisms. However these tests remain to be validated in a clinical setting.

The goal of the current study is to evaluate the diagnostic value of plasma detection of bacterial DNA in ICU patients with a clinical suspicion of bacterial infection.

DETAILED DESCRIPTION:
The goal of the current study is to evaluate the diagnostic value of plasma detection of bacterial DNA in ICU patients with a clinical suspicion of bacterial infection.

Definitions of septic syndromes based from the ACCP/SCCM expert panel. Terms Definition criteria Infection Invasion by microorganisms of an normally sterile tissue

Systemic inflammatory response Syndrome (SIRS) At least 2 of 4 following criteria:

* Temperature > 38°C or < 36°C
* Heart Rate > 90 beat/min
* Tachypnea > 20/min or PaCO2 < 32 mmHg
* WBC count > 12 000/mm3 or < 4 000/mm3 Sepsis SIRS related to an infectious process

Severe Sepsis Sepsis with :

* Arterial hypotension (SBP<90 mmHg, MAP<70 or SBP decrease < 40 mmHg)
* Or any other organ dysfunction :
* PaO2/FiO2 < 250 (or < 200 if pneumonia)
* Oliguria (< 0,5 ml/kg/h for at least 2 hours)
* Hyperlactacidemia ( > 3mmol/l)
* Platelet count < 80000/mm3 Septic shock Severe sepsis with persisting hypotension ( > 1 hour) despite adequate fluid resuscitation and requiring vasopressor support (epinephrine or norepinephrine).

SBP: Systemic blood pressure, MAP: Mean arterial blood pressure,

All codes and definitions are established prior to study initiation. The following information are recorded: age and sex, admission category (medical, scheduled surgery, or unscheduled surgery), origin (home, ward, or emergency room), and McCabe score, ICU and hospital mortality. Severity of illness was evaluated on the first ICU day using the Simplified Acute Physiology Score (SAPS II), Sepsis-related Organ Failure Assessment (SOFA) score, and Acute Physiologic and Chronic Health Evaluation (APACHE) II score. Knaus scale definitions were used to record preexisting chronic organ failures including respiratory, cardiac, hepatic, renal, and immune system failure.

The presence or absence of infections was documented according to the standard definitions developed by the Centers for Disease Control; We will determine three groups: 1. patients with documented infection 2. patients without documented infection and 3. patients with suspected but non documented infection.

Study protocol Four centers will participate (65 beds overall). Along with clinical C-reactive protein (CRP) and procalcitonin (PCT) measurements used in clinical routine lab measurements, two blood samples (4.5 mL each) will be collected. CRP and PCT are collected routinely when patient meet criteria for SIRS in all three ICUs to helps us distinguishing infectious from non-infectious SIRS. One whole blood on EDTA will be rapidly processed for bacterial/fungi DNA detection. (frozen until analysis or within 72 hours the sample kept at 4°C).

The second sample using tubes containing Gel and dipotassium EDTA allowing separation after centrifugation (1500g for 10 minutes at 4°C) of the plasma from (white and red) blood cells without any manipulation and thus lowering risk any nurses' occupational exposure. Then the plasma will be stored at -80°C until analysis. Blood collection will be performed when SIRS criteria will be met either at admission or later on during the ICU stay (suspicion of surperinfection).

Bacterial and Fungal DNA detection The bacterial and Fungal DNA detection will be performed using the Multiplex PCR pathogen detection VYOOTM (SIRS-Lab GmbH, Jena, Germany). VYOOâ combines culture-independent pathogen-derived nucleic acids concentration and multiplex PCR-based species detection. The multiplex PCR delivers results of high therapeutic value within ~6 hours and detects 34 bacterial and 6 fungal species that cause life-threatening infections as well as five most frequent resistance markers. In order to ensure highest clinical validity, the primer selection of the species and the antibiotic resistances bases on international study results on septic infections. The system was proved to be far less susceptible for contaminations than blood cultures or alternative NAT protocols and ensures increased specificity and sensitivity.

VYOOâ achieves its high sensitivity with the included sample preparation system LOOXSTER® which bases on SIRS-Lab's proprietary PUREPROVE® technology. LOOXSTER® specifically concentrates the minute quantity of bacterial and fungal DNA from a huge human DNA background. Total DNA is applied onto an affinity chromatography column with a matrix-immobilized DNA binding protein that recognizes definite motives within the pathogen DNA. More than 90% of the human background DNA is removed. This effect substantially increases the sensitivity of the downstream multiplex PCR protocol and simultaneously reduces the time-to-result.

The pathogen cells within 5 ml whole blood are disrupted mechanically using glass beads (0.1/2.5 mm in diameter) and a lysis device (e. g. FastPrep®-24, MP Biomedicals, Solon, OH, USA). After a proteolytic digestion step, total DNA is isolated using a short spin column protocol. The total DNA is dissolved in an appropriate buffer and applied to the LOOXSTER® spin column. The final bacterial plus fungal/human DNA ratio is significantly increased and the concentrated pathogen DNA is directly used for multiplex PCR. Generated pathogen specific amplicons are visualized by gel electrophoresis and compared with VYOOâ-specific DNA length markers for the proof of present pathogens or resistances. An alternative amplicon attribution is achieved by hybridization (ATâ system, Clondiag), which ensures a higher degree of specificity and sensitivity.

Cytokines detection by ELISA Dosage of plasma cytokines (IL-6, 8, 10) will be performed by ELISA methods using commercially available kits (R&D systems, Minneapolis, MN) or by Bio-Plex Multiplex Cytokine Assay (BioRad Lab., Hercules, CA).

Endotoxin & Peptidoglycan detection For endotoxin dosage, we used Limulus Amebocyte Lysate (LAL) reagent water (LRW) (Biowhittaker) and non-pyrogenic pipettes and tips (Costar). The samples will be diluted with LRW in non-pyrogenic 96-well culture plates (Costar). Blood samples will be collected in endotoxin free tubes containing a gel that after centrifugation makes a barrier between the cellular pellet and the plasma (Becton Dickinson, Franklin Lakes, NJ). The plasma will be then transferred to non-pyrogenic tubes and kept at -20°C until tested. Detection of bacterial endotoxin in plasma is hindered by its yellow coloration that interferes with the Limulus amebocyte lysate test and gives an absorbance at 405 nm, but also by the presence of inhibitors. We overcame the background absorbance of plasma using a Diazo-coupling Limulus amebocyte lysate assay that gives a magenta coloration (Associates of Cape Cod Inc.). Furthermore, in order to inactivate the inhibitors, plasma were diluted 1:4 in LRW and heated for 30 min at 60°C as it has been shown that this dilution and heating procedure allow optimal endotoxin detection in plasma. After heating, 50 μl of diluted plasma were transferred in 96-well culture plate and incubated with the same volume of Limulus amebocyte lysate for 30 min at 37°C. The reaction will be stopped, as specified by the manufacturer, by successive addition of 50 μl of sodium nitrite in HCl, 50 μl of ammonium sulfamate and 50 μl of N-(1-naphthyl)-ethylenediamine (NEDA) that form a diazotized magenta derivative. The optical density will be read at 570 nm and endotoxin concentration will be determined by comparison with an endotoxin standard curve. The detection limit of the test is 0.02 EU/ml of endotoxin.

Peptidoglycan will be measured according to a newly experimental procedure set up in Dr. Cavaillon's laboratory. The technique that detects peptidoglycan from both Gram-positive and Gram-negative bacteria has already been shown to detect peptidoglycan in plasma from patients with sepsis. Because a patent has been applied no further technical information can be presently provided in the present version but will be added as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* At least SIRS criteria at admission or during ICU stay.

Exclusion Criteria:

* age <18 year old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ICU patients older than 18 years old, with a SIRS, severe sepsis or septic shock will be included in this cohort study.
  SIRS, Severe sepsis and shock septic will be defined according to the definition used by a panel of experts from the American College of Chest Physicians/Society of Critical Care Medicine
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Using PCR we will determine the accuracy of these tests in identifying bacteria or fungi responsible of the infection. | End of the ICU stay

SECONDARY OUTCOMES:
We will examine whether or not cytokines' profile, levels of endotoxin and peptidoglycan help to discriminate infectious from non-infectious SIRS. | The assays will be done later on (within 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Adrie, MD, Principal Investigator — Delafontaine Hospital; Mehran Monchi, MD, Study Director — Jacques Cartier Institute
Locations (5):
- France (5):
  - Jacques Cartier Institute, Massy
  - Saint louis Hospital, Paris
  - Saint Joseph Hospital, Paris
  - Pasteur Institute, Paris
  - Delafontaine Hospital, Saint-Denis